CLINICAL TRIAL: NCT01614548
Title: Comparisons of Management and Outcome of Prostate Cancer in Central China Between 2003 and 2008: A Multi-institutional Report
Brief Title: Management of Prostate Cancer in Central China
Status: Completed | Type: Observational
Sponsor: Zhengzhou University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); the cancer hospital of Zhengzhou University (Unknown); Third Affiliated Hospital of Zhengzhou University (Other); People's Hospital of Zhengzhou University (Other); Xinyang Central Hospital (Other); Zhoukou Central Hospital (Other); Center hospital of Nanyang (Unknown); Center hospital of Shangqiu (Unknown); Zhumadian Central Hospital (Other); Anyang Regional Hospital (Other); Luoyang Central Hospital (Other); First People's Hospital of Kaifeng (Other)
Responsible Party: Principal Investigator, Liu Bingqian, Principal Investigator, Zhengzhou University
Other Study IDs: ZZU2012
Record Dates: First submitted 2012-06-02; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: Prostatic Neoplasms; Prostate Cancer; Disease Management; Rural; Urban
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all patients: We selected 9 cities (Zhengzhou, Luoyang, Kaifeng, Anyang, Xinyang, Zhoukou, Shangqiu, Nanyang, Zhumadian) by probability proportional to size sampling from geographical regions in central China. All cases with complete follow-up data of histological-proven prostate cancer treated in 2003 and 2008 at 14 department of urology in the 9 cities were retrospectively collected. Only patients with newly diagnosed prostate cancer were included in the study. Those with a history of prostate cancer who were treated for another disease were excluded from study.

SUMMARY:
Some recent reports indicate that incidence of prostate cancer is increasing rapidly in China. However, no large-scale survey of prostate cancer has been done in central China, few data are available regarding its management. The investigators aimed to analyze the management of prostate cancer and compare the outcome of patients with such a survey.

The investigators collected data of patients diagnosed with prostate cancer from the 2003 and 2008 in central China. Data were disaggregated by rural and urban hukou. The survival rate of patients was analyzed using Kaplan-Meier method. Prognostic factors were analyzed using the log-rank test and Cox proportional hazards model.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed prostate cancer were included in the study. Exclusion Criteria:
* Those with a history of prostate cancer who were treated for another disease were excluded from study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all inpatients with prostate cancer in 14 hospitals
Sampling Method: Probability Sample
Enrollment: 789 (Actual)
Dates: Start 2003-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 years
  overall survival that was defined as the interval from the date of diagnosis to the Medicare date of death

CONTACTS AND LOCATIONS:
Overall Officials: Liu Bingqian, Ph.D MD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- the first affiliated hospital of Zhengzhou University, Zhengzhou, Henan, China